CLINICAL TRIAL: NCT05814120
Title: Chang Gung University of Science and Technology
Brief Title: Effectiveness of Basic Life Support Training for Rural Community Dwelling Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University of Science and Technology (Other)
Responsible Party: Principal Investigator, Ching-Ching Su, Assistant Professor, Chang Gung University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 201600580B0
Record Dates: First submitted 2023-01-31; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Community Dwelling
Keywords: Basic Life Support; Rural Community Dwelling; Elderly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Geriatric-specific BLS training program
  Interventions: Behavioral: BLS training program

INTERVENTIONS:
Behavioral: BLS training program — BLS training program was in accordance with the 2020 AHA cardiopulmonary resuscitation (CPR) guidelines. The BLS training program adopts 4D teaching techniques, namely description (Describe), demonstration (Demo), implementation (Do), feedback (Debriefing).

SUMMARY:
The goal of this pre-post study is to test the effectiveness of basic life support (BLS) training for rural community-dwelling Elderly. The main question it aims to answer are can the training program tailored for rural elderly improve basic life support knowledge, attitude, and skills? Participants will receive an innovative BLS training program.

ELIGIBILITY:
Inclusion Criteria:

age older than 65-year-old, intact cognition, coordinated activities, and no history of severe cardiovascular disease, asthma, or lower extremity impairment.

Exclusion Criteria:

severe visual and hearing impairment, impractical to move, and mental illness.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 218 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Changes to the BLS Knowledge Questionnaire | Completion by study, average 60 minutes.
  The BLS knowledge assessment consisted of 10 questions with structured "yes" or "no" answers and was based on expert consensus from the AHA (AHA, 2020). Scores were calculated based on the number of correct answers given, with higher scores indicating a greater understanding of BLS.
Changes to the BLS attitude Questionnaire | Completion by study, average 60 minutes.
  The BLS attitude questionnaire contained five statements with five-point Likert-type scale responses ranging from "strongly agree" to "strongly disagree." Positive attitudinal answers awarded higher scores.
The observable BLS skill checklist | Completion by study, average 60 minutes.
  The observable BLS skill checklist included ten steps related to BLS practices, such as assessing responsiveness, calling for help, and using an AED. The researcher completed the checklist and rated each step on a 2-point scale, with higher scores indicating better BLS practices.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University of Science and Technology, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: No